CLINICAL TRIAL: NCT06646237
Title: Liquid Biopsy by Measuring Pleural Fluid Mycobacterium Tuberculosis Cell-free DNA (MTB cfDNA) Level to Diagnose Tuberculous Pleuritis in a Real-world Setting
Brief Title: Diagnostic Utility of Mycobacterium Tuberculosis Cell-free DNA in Hong Kong
Acronym: MYDNITE-3
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: MYDNITE-3
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis, Pleural; Pleural Biopsy
Keywords: Tuberculous pleuritis; cell-free DNA; Tuberculosis; pleural biopsy
MeSH Terms: conditions — Tuberculosis, Pleural; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Pleural fluid and blood obtained from patients with TBP and non-TBP will be stored for subsequent genetic sequencing techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBP: Patients with definite or probable tuberculous pleuritis
- Non-TBP: Patients without tuberculous pleuritis

SUMMARY:
Tuberculosis (TB) is an endemic infectious disease in Hong Kong and a global health threat. Tuberculous pleuritis (TBP) is the most common form of extrapulmonary tuberculosis in China. Its presentation is frequently non-specific and the diagnosis is challenging due to its paucibacillary nature. Various studies have shown that there are limitations for conventional diagnostic modalities, including low sensitivity for pleural fluid microbiological tests (acid-fast bacilli [AFB] stain, Mycobacterium tuberculosis [MTB] culture and MTB polymerase chain reaction [PCR]), lack of specificity for pleural fluid biomarkers (adenosine deaminase) especially in low TB prevalence regions, invasiveness for pleural biopsy (AFB stain, MTB culture and MTB PCR by bedside or pleuroscopy biopsy). The diagnostic journey can be lengthy due to the long turnaround time for microbiological tests and the need for multiple invasive diagnostic procedures. Therefore, the diagnosis of TBP is frequently based on a composite of clinical, radiological and laboratory endpoints to maximise the diagnostic yield and limit the invasiveness.

The application of pleural fluid MTB cell-free DNA (cfDNA) as a liquid biopsy to diagnose tuberculous pleuritis has been explored. Previous study groups focused on TB-specific single gene fragments revealed diagnostic sensitivity between 41.4% and 79.5%. Due to the suboptimal sensitivity, the clinical utility based on the previous technique was limited. Our study group has developed a novel MTB cfDNA assay based on different cfDNA processing techniques and interpretation algorithms, with sensitivity and specificity greater than 95% in diagnosing TBP. Since the performance of this novel MTB cfDNA assay was developed based on a limited number of selected cases, its clinical utility should be examined in a non-selective cohort of new-onset unilateral pleural effusion. Successful validation of MTB cfDNA in pleural fluid, as a liquid biopsy obtained through thoracentesis, can obviate the need to perform a pleural biopsy.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a key infectious disease burden globally. According to the Global TB Report by the World Health Organization (WHO) in 2023, Over seven million people were infected with TB in 2022, and 1.3 million died from the disease. China is among the top three countries with the highest TB burden, while Hong Kong has an intermediate burden of TB, with an average of 4,000 new cases per year.

TB infection can cause disease of various manifestations outside the lung parenchyma in about 25% of patients (extrapulmonary TB, EPTB), and is associated with worse treatment outcomes than pulmonary TB. Tuberculous pleuritis (TBP) is its most prevalent form in Hong Kong and China (41% to 50% of all EPTB). Although TBP can present with acute to subacute occurrence of unilateral pleural effusion, breathlessness and fever, its presentation is frequently non-specific. Due to its clinical and epidemiological importance, accurately discriminating TBP from other types of pleural effusion is crucial to shorten the diagnostic process and optimise the outcomes for these patients.

Laboratory challenges for diagnosing TBP Diagnosing TBP is challenging as the disease is caused by a small number of bacteria (paucibacillary nature) in the pleural space, which limits the diagnostic performance of various conventional diagnostic modalities. These limitations include low sensitivity for pleural fluid microbiological tests (acid-fast bacilli [AFB] stain, Mycobacterium tuberculosis [MTB] culture and MTB polymerase chain reaction [PCR]) and lack of specificity for pleural fluid biomarkers (adenosine deaminase [ADA]) especially in low TB prevalence regions. Although the yields of MTB culture and PCR on pleural tissue are higher, pleural biopsy (by bedside procedure or pleuroscopy) carries invasiveness and requires an additional procedure. Currently, no ideal test can achieve multiple diagnostic goals simultaneously, including high detection sensitivity, high specificity to exclude other diseases, short turnaround time, low invasiveness and detection of drug resistance. The diagnosis of TBP is practically based on a composite of clinical, radiological and laboratory endpoints. The diagnosis may occasionally be established clinically without any microbiological or histological proof (probable TBP).

Consequences of delayed TBP diagnosis The key clinical drawbacks of difficulty in diagnosing TBP include unnecessary invasive pleural interventions and delayed initiation of curative treatment. Our internal audit recently revealed that the initiation of treatment was delayed while waiting for confirmatory test results, and patients required a median of one additional procedure to establish the diagnosis, which included pleural biopsy with a more invasive nature. These patients had long hospital stays for workups and trials of multiple antibiotics for unresolved fever. Some patients may instead receive empirical anti-TB treatment based on compatible clinical presentations without confirmatory diagnostic investigation results. However, this is not without risk (e.g. hepatotoxicity), particularly in the elderly, who are more susceptible to TBP. A better diagnostic tool for TBP would mitigate these clinical challenges.

Liquid biopsy in pleural effusion: latest development from our group Liquid biopsy by detecting the cell-free DNA (cfDNA) in body fluids is a potential solution. When TB bacteria die or break down, the DNA fragments shed into the pleural space, forming Mycobacterium tuberculosis cfDNA (MTB cfDNA). Detecting the MTB cfDNA in the pleural fluid can directly prove the presence of TB bacilli or their subunits in the pleural space, which is an appealing option. Previous studies had employed MTB cfDNA to diagnose TBP, but the performance was variable. Che et al first measured MTB cfDNA by detecting the IS6110 insertion sequence. The sensitivity of diagnosing TBP was 75.0% (95% confidence intervals [CI] 63.7-86.3%) with specificity at 100.0% (95% CI 100.0-100.0%), and pleural fluid MTB culture-negative cases was included in the TBP group. The diagnostic sensitivity of MTB cfDNA was better than pleural fluid ADA, MTB culture and MTB PCR by Xpert MTB/RIF. Yang et al employed the same laboratory technique and found a high diagnostic sensitivity at 96.6% (95% CI 92.0-100.0%) in TBP cases defined by pleural fluid MTB or PCR positive status. However, the diagnostic sensitivity dropped to 79.5% (95% CI 72.4-86.7%) if pleural fluid MTB culture or PCR-negative cases were included in the TBP group. Similar findings were also reported by Sharma et al. All these study results reflected the heterogeneous diagnostic performance of MTB cfDNA. A negative pleural fluid MTB culture or PCR status, signifying a low bacterial load, can impair the clinical utility of MTB cfDNA.

Our group has recently developed a new laboratory assay measuring the MTB cfDNA levels, involving targeted sequencing through a capture-probe system and novel bioinformatics algorithm. The diagnostic performance remained robust even though pleural fluid MTB culture-negative cases were included, which can potentially obviate another invasive diagnostic procedure.

Need for a validation cohort before introducing to clinical practice Since the development cohort only contains a limited number of pleural fluid samples with definitive diagnoses, the true diagnostic accuracy of the novel MTB cfDNA assay can only be determined in a prospective, non-selective cohort reflecting the real-world situation, which will give a realistic diagnostic performance. This will confirm the clinical utility of MTB cfDNA assay before being introduced in clinical practice. We hypothesise that the novel MTB cfDNA assay remains robust in a prospective cohort and outperforms previously reported methods in discriminating pleural effusions due to TBP from non-TBP.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised for new-onset unilateral pleural effusion.
* Thoracentesis will be performed for pleural fluid analysis.
* Age equals or is above 18 years old
* Written informed consent is obtained

Exclusion Criteria:

* History of intrapleural therapy (including talc and fibrinolytic), surgical decortication or surgical pleurodesis in the ipsilateral pleural space in the past 3 months
* Concomitant use of at least two anti-TB medications (including isoniazid, rifampicin, pyrazinamide, ethambutol, amikacin, streptomycin, levofloxacin, moxifloxacin, linezolid) for more than consecutive 7 days in the past 3 months
* Failed to obtain informed consent due to patient's refusal or cognitive impairment.
* History of TBP in the ipsilateral pleural space
* Expected survival of less than three months from a different pathology (e.g. advanced metastatic malignancy) as that further pleural investigations may not be able to carry out if negative initial workup.
* Use of agents under research or not registered in the 30 days prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with definite or probably TBP will be recruited as positive control. Patients without TBP will be recruited as negative control.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of MTB cfDNA assay | 12 months
  The diagnostic performance (sensitivity and specificity) of MTB cfDNA assay with a pre-defined cutoff level in discriminating TBP and non-TBP in a prospective non-selective cohort of new-onset unilateral pleural effusions

SECONDARY OUTCOMES:
Factor affecting the test performance of MTB cfDNA assay | 12 months
  To compare the diagnostic performance of the MTB cfDNA assay in patients with different pleural fluid MTB culture status (positive or negative).
Compare the diagnostic performance | 12 months
  To compare the diagnostic performance of MTB cfDNA at pre-defined cutoff level (2 RP10M) with other diagnostic methods (pleural fluid ADA level, MTB culture, MTB PCR)
Estimate the proportion of pleural biopsy can be avoided | 12 months
  To estimate the potential reduction in pleural biopsies using a standardised biopsy indication rule compared to actual clinical practice, with sensitivity analyses for clinician variability, by the targeted sequencing-based MTB cfDNA assay. If the performance of MTB cfDNA assay is near perfect, pleural biopsy can be avoided in virtually all patients with suspected TBP. Alternatively, if the MTB cfDNA assay still misses some patients, the study will identify factors associated with false-negative results to guide when a pleural biopsy should be performed

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Study Director — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No